CLINICAL TRIAL: NCT02600091
Title: Exploring the Effectiveness of Mindfulness-based Cognitive Therapy to Improve Emotional Wellbeing and Glycaemic Control Among Adults With Diabetes
Brief Title: Mindfulness-based Cognitive Therapy to Improve Emotional Wellbeing and Glycaemic Control in Diabetes
Acronym: MILESTONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government); University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG12976-10
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2017-10

CONDITIONS: Anxiety; Depression; Diabetes
Keywords: Anxiety; Depression; Type 1 Diabetes; Mindfulness-based Cognitive Therapy; Glycaemic control
MeSH Terms: conditions — Anxiety Disorders; Depression; Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBCT Intervention (Experimental): Participants in the Mindfulness-based Cognitive Therapy Intervention arm will receive an 8-week programme in mindfulness-based cognitive therapy
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Waiting List Control (No Intervention): The participants who are allocated to the waiting list control group will receive usual care. They will receive the MBCT intervention 3 months after the intervention group complete their MBCT programme.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — The MBCT intervention is manualised and delivered to groups. The aim of the MBCT intervention is to increase mindfulness skills and to facilitate their use in relation to emotional wellbeing and diabetes self-management. Participants will attend on 8 occasions, once per week, for 2 hours. These meetings will have a standard structure. First, participants will describe their efforts to practice mindfulness at home over the previous week, followed by discussion of an educational topic relevant to the aims of the course. Finally, the group will do a mindfulness practice together, and the home practice for the following week will be set. In-between meetings, participants are asked to practice mindfulness by listening to an audio file or CD for about 30 minutes per day.
  Other Names: MBCT
  Arms: MBCT Intervention

SUMMARY:
Type 1 and 2 diabetes are challenging conditions to manage. Anxiety and depression are common among this group and are associated with poorer diabetes control. No trials have been conducted to ascertain the effectiveness of psychological interventions designed to alleviate significant levels of anxiety and/or depression and improve glycaemic control among those with diabetes who have significant difficulties with their emotional wellbeing and diabetes control.

The aim of this project is to establish if it is feasible to run a multi-site randomised controlled trial in Scotland exploring whether an 8-week mindfulness and self-management based intervention programme decreases anxiety and/or depression, and improves diabetes control. This feasibility study, based on the MRC framework for assessing feasibility and piloting methods, will assess the relative strengths and weaknesses of the intervention and study design, and pave the way for a larger and definitive trial.

DETAILED DESCRIPTION:
This is a feasibility trial informed by the MRC guidelines. It is a small RCT, where participants are randomised to either the MBCT intervention or waiting list control. Participants will be receiving their diabetes care in Aberdeen and Glasgow, and randomisation will occur at each site. The participants who are allocated to the waiting list control group will receive the MBCT intervention 3 months after the intervention group complete their MBCT programme.

The investigators will recruit participants using posters and leaflets, word of mouth from diabetes professionals, and from writing to those who are eligible. All of these methods are simply to raise awareness of the study. The intervention requires considerable commitment from participants (as indicated below) and this will be fully explained and explored. It will be up to potential participants to make initial contact with the research team, at which point they will be invited to the diabetes outpatient clinic for a discussion about what the project entails, the nature of mindfulness, and to go through the usual consent procedure.

In the cases of those people who agree to participate, the investigators will write to their GP and to their diabetes consultant to let them know that their patient has enrolled in the study, and provide brief information about the project.

The MBCT intervention is manualised and delivered to groups. The aim of the MBCT intervention is to increase mindfulness skills and to facilitate their use in relation to emotional wellbeing and diabetes self-management. Participants will attend on 8 occasions, once per week, for 2 hours. These meetings will have a standard structure. First, participants will describe their efforts to practice mindfulness at home over the previous week, followed by discussion of an educational topic relevant to the aims of the course. Finally, the group will do a mindfulness practice together, and the home practice for the following week will be set. In-between meetings, participants are asked to practice mindfulness by listening to an audio file or CD for about 30 minutes per day.

The research assistants will administer brief, self-report inventories at baseline; post-treatment and at 3 months follow-up to establish participants' level of mindfulness (Cognitive and Affective Mindfulness Scale-Revised);

1. diabetes-specific distress (Problem Areas in Diabetes; PAID);
2. anxiety and depression (Hospital Anxiety and Depression Scale; HADS);
3. positive emotional wellbeing (Warwick-Edinburgh Mental Wellbeing Scale);
4. satisfaction with treatment provision (Diabetes Treatment Satisfaction Questionnaire);
5. health-related quality of life (EQ-5D-5L),
6. and the Fear of Hypoglycaemia Scale.
7. During the intervention, the investigators will also ask participants to keep a diary of the number of times they completed the formal mindfulness exercises or these will be recorded using an specially designed app, and keep a record of attendance at group sessions.

Moreover, the investigators will request details of the frequency of severe hypoglycaemia (defined as occasion they needed help to correct blood glucose levels); mild-moderate (self-corrected) hypoglycaemia, and the number of admissions for diabetic ketoacidosis in the 6 months preceding the beginning of the MBCT course and for the period between the end of treatment and follow-up. The investigators will record the baseline HbA1c values and again obtain this at the 3 month follow-up point. Finally, participants will be asked to keep a diary of their health care use (for example, GP visits; calls to the diabetes specialist nurses; visits to secondary care diabetes health professional, and so on) during the previous 6 months at baseline and 3 months prior to follow-up. In addition, NHS Scotland; NHS Grampian, and NHS Glasgow electronic systems (eg, SCI-Diabetes and SCI-Store) will be used to obtain an accurate account of contact with secondary health professions.

The research assistants will also conduct one-to-one qualitative interviews with 10-15 participants, with equal numbers (for example, 6) from the MBCT group about 1 month after the end of the intervention. Interviews will be conducted with participants located in Aberdeen and Glasgow. These semi-structured interviews will focus on patients' views on why they volunteered; their expectations of the intervention; the acceptability of the intervention and measures; perceived benefits, and any difficulties they experienced during their participation. The investigators will also be keen to hear their thoughts on key characteristics of the facilitators; how best to attract potential participants in a future definitive trial, and ways to overcome any pragmatic difficulties, they experienced. The investigators will also attempt to contact all study drop-outs for a brief (5-10 minute) telephone interview on reasons for drop-out. This will include those who drop out prior to participation in the groups, those who drop out during group sessions, and those who complete group participation but fail to complete follow-up measures. Consent to contact for this reason will be obtained on entry to the study and this has proved acceptable in a current MBCT feasibility study using volunteer recruits. Analysis of qualitative data will be theoretically informed by Normalisation Process Theory (NPT) which specifically addresses the identification of barriers and facilitators to up-take of interventions or processes of change.

Standard demographic information including socio-economic status will be collected as will the co-existence of other conditions (co-morbidity). The investigators will also record standard diabetes health information such as time since diagnosis; any complications present, and any changes in medication between baseline and follow-up. The Scottish Index of Multiple Deprivation (SIMD) will be ascertained from participants' postcodes. The study will end on the date that the last data are collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over the age of 18 years)
* Type 1 or Type 2 diabetes, diagnosed at least 1 year ago
* Mild to moderate levels of anxiety and/or depression (ie, HADS scores of ≥ 8)
* Most recent HbA1c value of ≥ 75 mmol/mol (Type 1) or ≥ 61 mmol/mol (Type 2).

Exclusion Criteria:

* Severe mental health problems (such as severe depression with suicidal ideation, psychosis, personality disorder)
* Terminal illness
* Inability to give informed consent in English
* Inability to understand written and spoken English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recruitment/Retention Rates | 20 months
  This study aims to establish if a large scale, definitive RCT of a specifically designed mindfulness-based group intervention, with self-management activation embedded within the programme structure, for adults with diabetes and significant emotional distress, is feasible, justified, and potentially cost-effective. The primary outcome, which will decide whether or not a full trial is feasible, will be based on rates of recruitment and retention of participants.

SECONDARY OUTCOMES:
Acceptability | 20 months
  A secondary outcome, which will also influence whether or not a full trial is feasible, will be based on qualitative data collected from participants about their experience of the intervention and of taking part in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Keen, PhD, Principal Investigator — NHS Grampian
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Background] Feldman GC, Hayes AM, Kumar SM, Greeson JM, Laurenceau JP. Mindfulness and emotion regulation: the development and initial validation of the Cognitive and Affective Mindfulness Scale-revised (CAMS-R) Journal of Psychopathology and Behavioral Assessment 29 (3): 177-190 , 2007
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Bradley C. The Diabetes Treatment Satisfaction Questionnaire: DTSQ. In Handbook of Psychology and Diabetes: A Guide to Psychological Measurement in Diabetes Reseacrh and Practice. Edited by Bradlet C, Chur, Switzerland: Harwood Academic Publishers. 1994
- [Background] EuroQuol Group. EQ-5D-5L User Guide. Available from http://www.euroqol.org/fileadmin/user_upload/Documenten/PDF/Folders_Flyers/EQ-5D-5L_UserGuide_2015.pdf. Last accessed November 2015
- [Background] Gonder-Frederick LA, Schmidt KM, Vajda KA, Greear ML, Singh H, Shepard JA, Cox DJ. Psychometric properties of the hypoglycemia fear survey-ii for adults with type 1 diabetes. Diabetes Care. 2011 Apr;34(4):801-6. doi: 10.2337/dc10-1343. Epub 2011 Feb 23. PMID 21346182